CLINICAL TRIAL: NCT07186582
Title: Verona Coronary Physiology Interventional Registry
Acronym: VR-CP
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Roberto Scarsini, MD, PhD, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: VR-CP
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease (IHD); Coronary Heart Disease (CHD)
Keywords: Coronary Physiology; Fractional Flow Reserve (FFR); Radial Wall Strain; Intermediate Coronary Stenosis; Functional Coronary Angiography; Murray's law quantitative flow ratio; angiographic microvascular resistance
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: The VR-CP study cohort includes consecutive adult patients (≥18 years) who underwent coronary angiography for suspected ischemic heart disease and had at least one coronary lesion assessed by fractional flow reserve (FFR) or angiography-derived FFR.
  Interventions: Diagnostic Test: Coronary physiology assessment using Fractional Flow Reserve (FFR) as per standard of care and angiography-derived FFR

INTERVENTIONS:
Diagnostic Test: Coronary physiology assessment using Fractional Flow Reserve (FFR) as per standard of care and angiography-derived FFR — Functional assessment of coronary lesions performed using invasive FFR or angiography-derived FFR during coronary angiography as part of routine clinical care. No active intervention or treatment is assigned by the study.

SUMMARY:
The Verona Coronary Physiology Interventional Registry (VR-CP) is an observational study that collects information on patients with suspected coronary artery disease who underwent coronary angiography with a functional assessment of coronary stenoses. These functional tests include fractional flow reserve (FFR) or angiography-derived FFR, which help physicians understand whether a narrowing in the coronary arteries is likely to reduce blood flow to the heart.

The main goal of the study is to investigate whether the functional severity of coronary lesions is associated with future cardiovascular events, such as heart attack, the need for repeat procedures, or cardiovascular death. Additional objectives are to compare invasive FFR with angiography-derived FFR, to evaluate how these values relate to angina symptoms, and to analyze differences between patients treated conservatively with medications and those treated with coronary interventions.

The study is retrospective and single-center, including approximately 1,000 patients who underwent coronary physiology testing between 2010 and 2024 at the University Hospital of Verona. Follow-up information is obtained through review of medical records, outpatient visits, or telephone contacts, and patients will be followed for up to 10 years.

By combining detailed coronary physiology data with long-term clinical outcomes, this registry aims to improve understanding of which patients are at higher risk and to guide future strategies for the diagnosis and treatment of coronary artery disease.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains one of the leading causes of morbidity and mortality worldwide. Conventional coronary angiography is limited because it shows the anatomy of the vessels but does not always reveal whether a narrowing truly reduces blood flow. To address this limitation, physiological indices such as fractional flow reserve (FFR) and angiography-derived FFR have been developed to provide a more accurate assessment of the functional severity of coronary stenoses.

The VR-CP registry is designed to evaluate the long-term prognostic value of these functional measurements. Patients who underwent coronary angiography with physiology testing at the University Hospital of Verona are included, and their angiographic data are linked to subsequent clinical outcomes. Follow-up information is collected through hospital records, outpatient visits, and telephone contacts, with a focus on major cardiovascular events and patient-reported angina status.

This study provides a unique opportunity to analyze a large, consecutive cohort over a long observation period. By correlating physiological lesion characteristics with outcomes such as myocardial infarction, target vessel revascularization, cardiovascular death, and quality-of-life measures, the registry aims to identify high-risk patient subgroups and refine treatment strategies.

The knowledge gained from this registry may contribute to more personalized decision-making in patients with CAD, improve the use of physiology in daily practice, and ultimately guide strategies for balancing conservative management versus invasive revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary angiography with functional assessment by FFR or angiography-derived FFR (index procedure)
* Willing and able to provide informed, written consent
* Age ≥ 18 years at the time of the index procedure

Exclusion Criteria

* Impossibility to obtain informed consent
* Age < 18 years at the time of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who underwent coronary angiography for suspected coronary artery disease with functional assessment (coronary physiology) performed from 2010 to 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Vessel-Oriented Composite Endpoint (VOCE) | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Composite of cardiac death, target vessel myocardial infarction, and ischemia-driven target vessel revascularization as adjudicated by an independent Clinical Events Committee (CEC) blinded to patient clinical data.

SECONDARY OUTCOMES:
Cardiovascular death | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Deaths attributed to cardiovascular causes, adjudicated according to ARC-2 definitions.
Target vessel-related myocardial infarction | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Myocardial infarction classified as related to the target vessel, defined by the 4th Universal Definition of MI.
Target vessel revascularization | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Any ischemia-driven percutaneous or surgical revascularization of the target vessel, based on symptoms, ischemia testing, or invasive physiology criteria.
Hospitalization for unstable angina | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Number and timing of hospital admissions due to unstable angina.
Angina status (Seattle Angina Questionnaire) | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Assessment of angina symptoms and quality of life using the validated Seattle Angina Questionnaire.
Number of prescribed antianginal medications | At 12 months, and every 12 months thereafter up to 10 years after index coronary angiography
  Count of antianginal drugs prescribed to each patient during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Scarsini, MD, PhD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona (AOUI); Simone Fezzi, MD, Study Chair — AOUI Verona; Flavio Ribichini, MD, Study Chair — AOUI Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona(AOUI), Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: Undecided
At present, it has not yet been decided whether individual participant data (IPD) from this observational study will be shared with external researchers. Decisions on data sharing will be made considering ethical, legal, and institutional requirements. If a plan to share IPD is established, appropriate procedures for data access and privacy protection will be implemented.

DOCUMENTS (1):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT07186582/Prot_000.pdf